CLINICAL TRIAL: NCT03832686
Title: Investigation of Two Swallowing Therapy Models During Radiation Therapy for Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Heather Starmer, Clinical Associate Professor and Director of the Head and Neck Cancer Speech and Swallowing Rehabilitation Center, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB-48015; ENT0070 (Other: OnCore); NCI-2019-04958 (Other: NCI)
Record Dates: First submitted 2019-01-28; First posted 2019-02-06 (Actual); Results first posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Head Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Coach App (Experimental): Participants in the experimental arm (Group A) will receive a comprehensive swallowing rehabilitation app. This study seeks to determine if a mobile application may enhance adherence to swallowing therapy in patients undergoing radiation therapy for head and neck cancer. No devices - outside of the Smartphone already owned by the participant - will be used in this study. Similarly, no drugs, biological materials, or other substances will be used.
  Interventions: Other: Virtual Coach
- Standard of Care (No Intervention): The paper group (Group B) will be given paper exercise logs to fill out Participants will be educated regarding potential radiation-related side effects and trained in the same series of swallowing exercises by the SLP. The paper log treatment group will serve as a standard treatment group. As adherence is a primary goal of the target intervention, paper logging will be necessary to determine relative adherence while minimizing reporting bias.

INTERVENTIONS:
Other: Virtual Coach — The smartphone application, tailored to patients with HNC, will monitor patient progress while also providing a direct line to health care providers should any questions or concerns arise concerning their treatment. The mobile application will also feature instructional videos that describe the swallowing exercises in detail, providing patients with another resource to help improve their overall rehabilitation experience. Finally, home practice reminders and prompts will be used to help patients integrate the exercises into their daily routine.
  Arms: Virtual Coach App

SUMMARY:
Vibrent Health is partnering with Stanford Cancer Center to conduct a randomized control trial (RCT) using mobile health technology to enhance adherence and improve swallowing outcomes in patients undergoing radiation therapy for head and neck cancer.

DETAILED DESCRIPTION:
Head and neck cancer (HNC) is the 6th most common type of cancer in the world and has recently seen a dramatic rise in the United States due to a rise in the incidence of oropharyngeal cancers related to the human papillomavirus (HPV) . The majority of patients diagnosed with HNC receive radiation therapy at some point in their treatment, either in the definitive or post-operative setting. Dysphagia is a common consequence of treatment for HNC, experienced by approximately 50% of patients treated with radiation therapy. Post-treatment dysphagia has been associated with increased risk of morbidity/mortality as well as well-recognized deterioration of quality of life. Performance of swallowing exercises during radiation significantly reduces dysphagia risk; however, patient adherence to swallowing exercises during radiation treatment is limited. Thus, poor adherence stands as a major obstacle to achieving the best swallowing outcomes. In response to this, a mobile health application was developed to directly address barriers cited by patients as reasons for non-adherence. The objective is to conduct a randomized controlled trial to test the impact of the mobile application on adherence to prophylactic swallowing therapy during radiation for HNC.

ELIGIBILITY:
Inclusion Criteria:

* Study subjects ≥ 18 years of age.
* Fluent English speaking subjects.
* Study subjects capable of providing informed consent.
* Patients with newly diagnosed non-metastatic head and neck cancer of the oral cavity, oropharynx, nasopharynx, hypopharynx, and larynx that require bilateral neck radiation. Individuals with unknown primary head and neck cancer with nodal disease necessitating bilateral radiation will also be included.
* Study subjects with a previously untreated head and neck cancer diagnosis requiring a definitive course of radiotherapy requiring a prescribed dose of 60Gy or greater.
* Study subjects who have either an Android or Apple iOS-based smartphone or tablet compatible with the Vibrent application.
* Study subjects who have access to a sufficient monthly data plan (approximately 200 MB/month), or Internet connection.

Exclusion Criteria:

* Non-English speaking, or incapable of providing informed consent.
* Lack of smartphone, tablet, or Internet connection.
* Inability to use the Vibrent application.
* Patients being treated for head and neck cancer who do not receive some form of primary, adjuvant, or neo-adjuvant radiation therapy will not be considered for the study.
* Patients with recurrent disease.
* Pregnant women.
* Individuals under the age of 18.
* Individuals with contraindications to radiation therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2023-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Starmer, Principal Investigator — Stanford Universiy
Locations (3):
- United States (3):
  - Stanford Cancer Institute, Palo Alto, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Starmer HM, Klein D, Montgomery A, Goldsmith T, McCarroll L, Richmon J, Christopher Holsinger F, Beadle B, Jain P. Head and Neck Virtual Coach: A Randomized Control Trial of Mobile Health as an Adjunct to Swallowing Therapy During Head and Neck Radiation. Dysphagia. 2023 Jun;38(3):847-855. doi: 10.1007/s00455-022-10506-5. Epub 2022 Aug 12. PMID 35960394

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 98 participants were screened, 91 participants were randomized to a study arm.
Groups:
- Virtual Coach App: Participants use a comprehensive swallowing rehabilitation app to determine if a mobile application may enhance adherence to swallowing therapy.
- Standard of Care: Participants are educated regarding potential radiation-related side effects and trained in the same series of swallowing exercises by the SLP and complete paper exercise logs.
Period: Overall Study
Arm/Group | Virtual Coach App | Standard of Care
Started | 44 | 47
Completed | 33 | 34
Not Completed | 11 | 13
Not completed — Lost to Follow-up | 6 | 9
Not completed — Discontinued Intervention | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Virtual Coach App | Standard of Care | Total
Number analyzed (Participants) | 44 | 47 | 91
Age, Continuous [Median (Full Range); unit: years] | 61 [24 to 76] | 62 [32 to 76] | 62 [24 to 76]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 39 | 40 | 79
  Unknown/Not Reported | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 40 | 46 | 86
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 38 | 44 | 82
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 44 | 47 | 91

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving at Least 50% Adherence to Swallowing Exercises
Description: Measure of overall adherence to prescribed exercise protocol, by treatment group and radiation week.
Time Frame: 7 weeks
Population: Participants with available data at each respective timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Coach App | Standard of Care
Number analyzed (Participants) | 38 | 40
Participants
  Week 1 | 18 | 17
  Week 2 | 19 | 16
  Week 3 | 15 | 13
  Week 4: number analyzed (Participants) | 38 | 39
  Week 4 | 15 | 12
  Week 5: number analyzed (Participants) | 38 | 39
  Week 5 | 9 | 9
  Week 6: number analyzed (Participants) | 38 | 39
  Week 6 | 9 | 10
  Week 7: number analyzed (Participants) | 38 | 39
  Week 7 | 6 | 4

2. Secondary Outcome: Patient Perceived Swallowing Impairment as Measured by the MD Anderson Dysphagia Inventory (MDADI)
Description: The MD Anderson Dysphagia Inventory (MDADI) was selected to capture and quantify the patient perception of swallowing dysfunction. It is a 20-item patient reported survey that measures the impact of dysphagia on patients with HNC. Each item is scored on a 5 point scale with 1=lower function and 5=higher function. Possible scores range from 20-100 with higher scores indicating more normal swallowing function.
Time Frame: 19 weeks
Population: Participants who completed the intervention and were blinded at consent.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Coach App | Standard of Care
Number analyzed (Participants) | 32 | 34
score on a scale | 75.66 (13.6) | 76.35 (17.1)
Statistical Analysis 1: Comparison: Virtual Coach App vs Standard of Care; Test type: Other; p = 0.86, Logistic Regression — A p-value of <0.05 would be considered statistically significant

3. Secondary Outcome: Diet Level as Defined by the Functional Oral Intake Scale (FOIS)
Description: Functional Oral Intake Scale (measure of diet restriction). Scores range from 1-7 where lower scores reflect more limited oral intake and higher scores reflect more normal diet levels.
Time Frame: 19 weeks
Population: Participants who completed the intervention and were blinded at consent.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Coach App | Standard of Care
Number analyzed (Participants) | 32 | 34
score on a scale | 6.06 (1.0) | 5.94 (1.5)
Statistical Analysis 1: Comparison: Virtual Coach App vs Standard of Care; Test type: Other; p = 0.69, Logistic Regression — A p-value of <0.05 would be considered statistically significant

4. Secondary Outcome: Diet Restrictions as Measured by the Performance Status Scale Head and Neck
Description: Performance Status Scale Head and Neck measures eating in public (range 0-100; higher number is indicative of better function), and normalcy of diet (range 0-100, higher number is indicative of more normal function)
Time Frame: 7 weeks
Population: Participants who completed the intervention and were blinded at consent.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Coach App | Standard of Care
Number analyzed (Participants) | 32 | 34
score on a scale
  Eating in Public | 90.15 (19.4) | 86.12 (25.9)
  Normalcy of Diet | 79.12 (7.2) | 76.94 (7.1)
Statistical Analysis 1: Comparison: Virtual Coach App vs Standard of Care; Comparison of Eating in Public Score; Test type: Other; p = 0.47, Logistic Regression — A p-value of <0.05 would be considered statistically significant
Statistical Analysis 2: Comparison: Virtual Coach App vs Standard of Care; Comparison of Normalcy of Diet score; Test type: Other; p = 0.73, Logistic Regression — A p-value of <0.05 would be considered statistically significant

5. Secondary Outcome: Physiological Oropharyngeal Swallowing Impairment as Measured by the Modified Barium Swallow Impairment Profile (MBS-ImP)
Description: The Modified Barium Swallow Impairment Profile is a tool designed to quantify degree of impairment on 13 individual physiologic components visualized during a modified barium swallow where higher numbers reflect greater dysfunction. Score range: 0-4 for each physiologic component. The maximum possible Oral score is 22 and the maximum possible pharyngeal score is 29.
Time Frame: 19 weeks
Population: Participants who completed the intervention and were blinded at consent.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Coach App | Standard of Care
Number analyzed (Participants) | 32 | 34
score on a scale
  MBSImP Oral | 3.9 (2.9) | 4.21 (2.5)
  MBSImP Pharyngeal | 9.33 (3.8) | 8.18 (3.9)
Statistical Analysis 1: Comparison: Virtual Coach App vs Standard of Care; Comparison of MBSImP Oral score; Test type: Other; p = 0.65, Logistic Regression — A p-value of <0.05 would be considered statistically significant
Statistical Analysis 2: Comparison: Virtual Coach App vs Standard of Care; Comparison of MBSImP Pharyngeal score; Test type: Other; p = 0.24, Logistic Regression — A p-value of <0.05 would be considered statistically significant

6. Secondary Outcome: Depth of Bolus Entry Into the Laryngeal Vestibule as Measured Using the Penetration-Aspiration Scale (PAS)
Description: The Penetration Aspiration Scale measures the presence and depth of food/liquid material entering the airway and patient response to that material. This scale ranges from 1-8 with higher numbers indicating more abnormal function.
Time Frame: 19 weeks
Population: Participants who completed the intervention and were blinded at consent.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Coach App | Standard of Care
Number analyzed (Participants) | 32 | 34
score on a scale | 2.76 (2.1) | 2.42 (1.7)
Statistical Analysis 1: Comparison: Virtual Coach App vs Standard of Care; Test type: Other; p = 0.53, Logistic Regression — A p-value of <0.05 would be considered statistically significant

7. Secondary Outcome: Severity of Impairment of Swallowing Safety and Efficiency as Measured Using the Dynamic Imaging Grade of Swallowing Toxicity (DIGEST) Scale
Description: Dynamic Imaging Grade of Swallowing Toxicity (DIGEST) rates the safety and efficiency of the swallow. Safety and efficiency are rated on a scale of 0-4 with higher numbers indicating more abnormality. This scale also includes an overall impairment score which takes into consideration the safety and efficiency grade.
Time Frame: 7 weeks
Population: Participants who completed the intervention and were blinded at consent.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Coach App | Standard of Care
Number analyzed (Participants) | 32 | 34
score on a scale | 0.97 (1.0) | 0.82 (0.8)
Statistical Analysis 1: Comparison: Virtual Coach App vs Standard of Care; Test type: Other; p = 0.50, Logistic Regression — A p-value of <0.05 would be considered statistically significant

ADVERSE EVENTS:
Time Frame: Up to 19 weeks
Description: Per protocol, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Virtual Coach App | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/86/NCT03832686/Prot_SAP_000.pdf